CLINICAL TRIAL: NCT00354120
Title: Randomized Study for Comparison of Reduced Intensity Conditioning Protocols Containing Either Thymoglobuline or Alemtuzumab in Patients Undergoing Allogeneic Transplant From Voluntary Unrelated Donors
Brief Title: Thymoglobuline Versus Alemtuzumab in Patients Undergoing Allogeneic Transplant
Acronym: GLOBAL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gruppo Italiano Trapianto di Midollo Osseo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT:2005-000805-68
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Acute Myeloblastic Leukemia; Lymphoblastic Leukemia; Myelodysplasia; Chronic Myeloid Leukemia; Myelofibrosis; Lympho-proliferative Diseases
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Primary Myelofibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Alentuzumab
  Interventions: Drug: Alentuzumab
- 2 (Active Comparator): Globulina antilinfocitaria
  Interventions: Drug: Globulina antilinfocitaria

INTERVENTIONS:
Drug: Alentuzumab — Alentuzumab
  Arms: 1
Drug: Globulina antilinfocitaria — Globulina antilinfocitaria
  Arms: 2

SUMMARY:
The purpose of this study is to compare Reduced Intensity Conditioning protocols containing either Thymoglobuline or Alemtuzumab in patients undergoing allogeneic transplant from voluntary unrelated donors.

DETAILED DESCRIPTION:
The reduction of intensity of conditioning is currently indicated for patients who cannot undergo standard myelo-ablation due to their age, comorbidities or type of pathology. Furthermore, the rationale to use RIC regimens is based on the observation that the infusion of alloreactive donor lymphocytes may yield to a graft versus tumour effect. However, in this kind of regimens the morbidity and TRM due to GvHD are still a concern and in vivo T-depletion is a necessary treatment. Both monoclonal (Alemtuzumab) and polyclonal T-depletion protocols carry risks and benefits. Benefits being a better prophylaxis for GvHD, and risks being an higher incidence of post-transplantation infections and relapse. At the moment, it is not clear which type of regimen, monoclonal or polyclonal, is better for the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Group 1: 55-65 yo patients suffering from Acute Myeloblastic and Lymphoblastic Leukemia, Myelo-displasia, Chronic Myeloid Leukemia and Idiopathic Myelofibrosis (according to IBMDR operative manual)
* Group 2: patients <= 65 yo suffering from lympho-proliferative diseases according the REAL classification:
* High-doses chemotherapy relapsed CLL (B and T)
* Follicular lymphoma relapsed after 2 standard chemotherapy regimens or after high-doses chemotherapy
* Mantellar lymphoma relapsed after 1 standard chemotherapy regimen or after high-doses chemotherapy
* Lympho-plasmacytoid and B marginal zone lymphoma in relapse after 2 standard chemotherapy regimens or after high-doses chemotherapy
* Advanced (stage ≥ III A) or relapsed T lymphomas
* Large B-cells lymphomas in 2nd or further complete remission after relapse from high dose chemotherapy and autotransplant or after 2 standard chemotherapy regimens
* Fungal mycosis in advanced stage (≥ III A) or in chemosensitive relapse after 2 lines of chemotherapy and Sezary syndrome in chemosensitive relapse after 1 line of chemotherapy
* Hodgkin disease relapse after autotransplant with chemosensitive disease or in relapse after 1 year from chemotherapy and not eligible for autotransplant since an insufficient mobilization of autologous hemopoietic stem cells.

Exclusion Criteria:

* Performance status < 70% (Karnofsky)
* Left ventricular cardiac ejection fraction < 40% or receiving treatment for heart failure
* DLCO pulmonary < 40% or receiving continuous oxygen therapy
* Neuropathy (previous or at present)
* Pregnancy
* Patients with arterial hypertension not controlled with multi-pharmacological treatments
* HIV positive
* B-CLL with clear evidence of transformation into Richter syndrome
* Mycosis fungoides with clear evidence of transformation into blasts
* Hodgkin's disease refractory to chemotherapy
* Absence of informed consent
* Psychiatric disease or other condition compromising the signing of the informed consent form or compliance with the treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2005-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 3 years
Event Free Survival and Disease Free Survival | 3 years
Safety: | 3 years
Major infective complications (CMV and EBV related PTLD) | 3 years
Acute and chronic GvHD | 3 years

SECONDARY OUTCOMES:
Haematological and immunologic reconstitution | 3 years
Incidence of CMV and EBV reactivation | 3 years
Other infective complications | 3 years
Other toxicities | 3 years
Need for DLI | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Rambaldi, MD, Study Chair — Divisione di Ematologia - Ospedali Riuniti di Bergamo
Locations (22):
- Italy (22):
  - Ematologia e Centro Trapianti Midollo Osseo - Ospedale IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - Divisione Ematologia - Ospedale "SS. Antonio, Biagio e Cesare Arrigo", Alessandria
  - Clinica di Ematologia - Ospedali Riuniti di Ancona, Ancona
  - Divisione di Ematologia - Ospedali Riuniti Bergamo, Bergamo
  - S.C. Ematologia - Azienda Ospedaliera S. Croce e Carle, Cuneo
  - Cattedra di Ematologia - Azienda Ospedaliera di Careggi, Florence
  - Trapianti Midollo Osseo - Div. di Ematologia 2 - Ospedale S. Martino, Genova
  - Divisione di Ematologia - Istituto Nazionale dei Tumori, Milan
  - U.O. Ematologia I - Centro Trapianti di Midollo - Ospedale Maggiore - Policlinico Mangiagalli e Regina Elena, Milan
  - Divisione Ematologia - Azienda Ospedaliera Universitaria - Policlinico -, Modena
  - Cattedra di Medicina Interna ed Ematologia - Ospedale S. Gerardo de' i Tintori - Università degli Studi di Milano, Monza
  - Divisione Ematologia con trapianto - Ospedale "V. Cervello", Palermo
  - Dipartimento di Ematologia - IRCCS Policlinico S. Matteo - Università di Pavia, Pavia
  - Dip. di Ematologia - Unità di Terapia Intensiva Ematologica per il Trapianto Emopoietico - Ospedale Civile di Pescara, Pescara
  - Ematologia - Ospedale S. Chiara, Pisa
  - Centro Unico Regionale Trapianti di Midollo Osseo - Ospedale Bianchi-Melacino-Morelli, Reggio Calabria
  - Cattedra di Ematologia - Università La Sapienza, Roma
  - Divisione di Ematologia - Istituto di Semeiotica Medica - Policlinico A. Gemelli, Roma
  - U.O. di Ematologia e Trapianti di Midollo Osseo - Azienda Osp. S. Camillo-Forlanini / Padiglione Morgagni, Roma
  - Dipartimento di Oncologia Medica ed Ematologia - Istituto Clinico Humanitas, Rozzano (MI)
  - Ematologia 2 - ASO San Giovanni Battista, Torino
  - Clinica Ematologica - Policlinico Universitario, Udine

REFERENCES:
- See also: GLOBAL Official Web Site — https://heart.negrisud.it/gitmo/default1.htm